CLINICAL TRIAL: NCT04949789
Title: A Randomized, Placebo-controlled, Blinded, Pilot Study to Evaluate Efficacy of Botanical Extracts as Protein Amplifier for Skeletal Muscle Strength & Growth.
Brief Title: Pilot Study to Evaluate Efficacy of Botanical Extracts as Protein Amplifier for Skeletal Muscle Strength & Growth.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: EB/200301/POLY/SMS
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2021-10

CONDITIONS: Muscle Strength
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Arm 1 (Placebo without Exercise) Arm 2 (Placebo with Exercise) Arm 3 (IP I) Arm 4 (IP II) Arm 5 (IP III)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo without Exercise (Other): 2 Capsules to be taken 30 minutes before breakfast.
  * Whey Protein (standardized for NLT 90% AA): 48 gms of Whey protein isolate (WPI) will be taken by participants daily in two divided doses of 24 gms dissolved in 200 ml of water with their breakfast and dinner.
  * On testing and exercise days, WPI with IP will be taken 30 mins prior to the exercise without breakfast consumption.
  Interventions: Other: Placebo without Exercise
- Placebo with Exercise (Other): 2 Capsules to be taken 30 minutes before breakfast.
  * Whey Protein (standardized for NLT 90% AA): 48 gms of Whey protein isolate (WPI) will be taken by participants daily in two divided doses of 24 gms dissolved in 200 ml of water with their breakfast and dinner.
  * On testing and exercise days, WPI with IP will be taken 30 mins prior to the exercise without breakfast consumption.
  Interventions: Other: Placebo with Exercise
- IP I (Other): 2 Capsules to be taken 30 minutes before breakfast.
  * Whey Protein (standardized for NLT 90% AA): 48 gms of Whey protein isolate (WPI) will be taken by participants daily in two divided doses of 24 gms dissolved in 200 ml of water with their breakfast and dinner.
  * On testing and exercise days, WPI with IP will be taken 30 mins prior to the exercise without breakfast consumption.
  Interventions: Other: IP I
- IP II (Other): 2 Capsules to be taken 30 minutes before breakfast.
  * Whey Protein (standardized for NLT 90% AA): 48 gms of Whey protein isolate (WPI) will be taken by participants daily in two divided doses of 24 gms dissolved in 200 ml of water with their breakfast and dinner.
  * On testing and exercise days, WPI with IP will be taken 30 mins prior to the exercise without breakfast consumption.
  Interventions: Other: IP II
- IP III (Other): 2 Capsules to be taken 30 minutes before breakfast.
  * Whey Protein (standardized for NLT 90% AA): 48 gms of Whey protein isolate (WPI) will be taken by participants daily in two divided doses of 24 gms dissolved in 200 ml of water with their breakfast and dinner.
  * On testing and exercise days, WPI with IP will be taken 30 mins prior to the exercise without breakfast consumption.
  Interventions: Other: IP III

INTERVENTIONS:
Other: Placebo without Exercise — 2 Capsules to be taken 30 minutes before breakfast.
  Arms: Placebo without Exercise
Other: Placebo with Exercise — 2 Capsules to be taken 30 minutes before breakfast.
  Arms: Placebo with Exercise
Other: IP I — 2 Capsules to be taken 30 minutes before breakfast.
  Arms: IP I
Other: IP II — 2 Capsules to be taken 30 minutes before breakfast.
  Arms: IP II
Other: IP III — 2 Capsules to be taken 30 minutes before breakfast.
  Arms: IP III

SUMMARY:
Sponsor proposes ingredients that when added to daily whey supplementation, can lead to increased muscle strength, improves sleep quality and reduction in fatigue level.

DETAILED DESCRIPTION:
The present study is a randomized, blinded, placebo-controlled, pilot study. Approximately 40 males aged between ≥ 20 and ≤ 35 years, will be screened. Each trial arm will have at least 5 completed after accounting for dropout/withdrawal rate of 20%. The treatment duration for all the study participants will be 28 to 56 days (Day 56 is only applicable for participants with less than 10% increase in weight leg pressed for 1 RM on Day 28. All participants in arm 1 of study will have their end of study visit on Day 28).Sponsor proposes ingredients that when added to daily whey supplementation, can lead to increased muscle strength, improves sleep quality and reduction in fatigue level.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 20 - 35 years with active lifestyle moderate physical activity level as per International Physical Activity Questionnaire.
2. Recreationally active but not participating in resistance type training on regular basis.
3. Body mass index (BMI) 22 - 29.9 kg/ m2
4. Participants with an Insomnia Severity Index score ≥7 and ≤14
5. Ready to refrain from caffeinated products and intense strength/ endurance exercise for 24 hrs. prior to the exercise lab visit.
6. Fasting Glucose ≤ 110 mg/ dl
7. Systolic Blood Pressure ≤ 129 mm Hg and Diastolic Blood Pressure ≤ 89 mm Hg
8. TSH (thyroid stimulating hormone) ≥0.4 and ≤ 4.9 mIU/L

Exclusion Criteria:

1. Engaged in structured weight training during the previous 12 months prior to screening.
2. Presence of chronic disease.
3. Changes in body weight more than 4.5 kg (10 pounds) in the past three months.
4. Participants with uncontrolled hypertension.
5. Participants who are diagnosed with Type II Diabetes Mellitus.
6. History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic, or neurologic disorders.
7. Allergy to whey or herbal ingredients.
8. Participants who have any other disease or condition, or are using any medication, that in the judgment of the investigator would put them at unacceptable risk for participation in the study or may interfere with evaluations in the study or noncompliance with treatment or visits.
9. Participants who have been part of a clinical trial within 90 days prior to the screening.
10. Participants who have used whey or other supplemental proteins anytime in last 3 months

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
1-Repetition Maximum | Day 0 to Day 28 and /or day56
  The final weight lifted successfully for atleast 1 repetition but could not complete 3 repetition will be recorded as 1- RM.
  Change in muscle strength as indicated by increase in 1Repetition Maximum leg press weight

SECONDARY OUTCOMES:
Body fat composition: Lean Muscle Mass by Dual-energy X-ray absorptiometry | Day 0 to Day 28 and /or day56
  Increase in lean muscle mass by DXA
Quality of Sleep: Modified Insomnia Severity Index | Day 0 to Day 28 and /or day56
  Improvement in sleep quality as assessed by the modified Insomnia Severity Index
Visual Analogue Scale for Fatigue | Day 0 to Day 28 and /or day56
  Reduction in fatigue level as assessed by the 11-point Visual Analogue scale for Fatigue
Mid-thigh Girth | Day 0 to Day 28 and /or day56
  Increase in mid-thigh muscle-girth (prior to exercise) at midpoint between inguinal fold and superior border of patella.
Digestive diary | Day 0 to Day 28 and /or day56
  Participants will be asked to fill out a paper/online digestive diary to monitor any significant changes that might occur to the digestive system due to the consumption of WPI and the IP.
  there should be No significant effect on digestive system as per participant digestive diary.

CONTACTS AND LOCATIONS:
Overall Officials: Dr, Anjali Jain, BHMS, Principal Investigator — Vedic lifesciences
Locations (1):
- Vedic Lifesciences, Mumbai, Maharashtra, India